CLINICAL TRIAL: NCT06184204
Title: Prospective, National, Multicentric, Observational Study to Evaluate the Safety, Efficacy and Quality of Life of Patients With Atrial Fibrillation, Treated With Trombix® (Rivaroxaban).
Brief Title: Observational Study:Safety,Efficacy and Quality of Life of Patients With Atrial Fibrillation, Treated With Trombix®
Acronym: TROMBIXDZ
Status: Completed | Type: Observational
Sponsor: Beker Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: TROMBIX.DZ _version 3
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
Keywords: real life; observational; safety; efficacy
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with confirmed diagnosis of Atrial fibrillation: male, female, 19 or more of age with confirmed diagnosis of Atrial fibrillation
  Interventions: Drug: Trombix® (Rivaroxaban)

INTERVENTIONS:
Drug: Trombix® (Rivaroxaban) — 20mg or 15 mg as per the doctor's prescription
  Other Names: Trombix®

SUMMARY:
The rational behind this observational study is to collect real life data about the use of Trombix® (Rivaroxaban) among patients with atrial fibrillation in Algeria . The aim is to evaluate the safety, efficacy and quality of life.

DETAILED DESCRIPTION:
Trombix® (Rivaroxaban) is used for the treatment of patients with atrial fibrillation. BEKER laboratories are conducting an observation study to evaluate its use among Algerian population in regards to its safety, efficacy and the quality of life of patients after its use.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged ≥ 19 years.
* Patient with a diagnosis of atrial fibrillation who requires treatment with Trombix® or switch of Anti-Vitamin K treatment toTrombix® (patient not balanced with current treatment or wishing to change treatment with better manageability).
* Patient being able to provide free and informed written consent before the study.

Exclusion Criteria:

* Hypersensitivity to the active ingredient or to one of the excipients indicated in the Summary of Product Characteristics of Trombix®
* Clinically significant progressive bleeding.
* Injury or illness, if considered to be at significant risk of major bleeding. This may include: current or recent gastrointestinal ulceration, presence of malignant tumors with a high risk of bleeding, recent brain, spinal or ophthalmic surgery, recent intracranial hemorrhage, known or suspected esophageal varices, arteriovenous malformations, vascular aneurysms or major intra-spinal or intracerebral vascular anomalies.
* Concomitant treatment with any other anticoagulant, for example, unfractionated heparin (UFH), low molecular weight heparins (enoxaparin, dalteparin, etc.), heparin derivatives (fondaparinux, etc.), oral anticoagulants (warfarin, dabigatran exilate, apixaban, etc.) except in specific circumstances of switching from anticoagulant treatment or in the case of administration of UFH at doses necessary to maintain the permeability of a central venous or arterial catheter.
* Liver injury associated with coagulopathy and clinically significant bleeding risk, including cirrhotic patients with Child Pugh score class B or C.
* Pregnancy and breast feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects in the study were enrolled from different centers (public and private sectors) across different regions in the country; East, Center and West of Algeria.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-06-22 (Actual)

PRIMARY OUTCOMES:
Assessment of reported Serious Adverse Effects linked to Trombix ® | 12 months
  * Assessment of serious adverse effects "major bleeding" linked to Trombix® reported as per the current medical practice for the following:
  * Incidence of intracranial hemorrhages
  * Incidence of hemorrhages requiring hospitalization with transfusion
  * Incidence of fatal hemorrhages
  * Incidence of critical organ bleeding
  * Incidence of gastrointestinal bleeding

SECONDARY OUTCOMES:
Epidemiological profile of patients: demographic data, pathological history, clinical profile at inclusion | 12 months
  Description the epidemiological characteristics of the patients: demographic data, pathological history, clinical profile at inclusion
Minor hemorrhages linked to Trombix® | 12 months
  Assessment of the Incidence of minor hemorrhages linked to Trombix® leading to definitive cessation of treatment
Incidence of any adverse effects | 12 months
  Assessment of the incidence rate of any adverse effects
Incidence of Trombix® treatment interruptions during 12 months of follow-up | 12 months
  Assessment of the percentage of patients who stopped Trombix® treatment during the 12 months of follow-up
Relative risk linked to each cause for stopping the treatment with Trombix® during follow-up | 12 months
  Identification of the causes behind stopping treatment with Trombix®
Incidence of severe thromboses: ischemic stroke / MI / non CNS-Systemic embolism | 12 months
  Assessment of the occurrence rate of ischemic stroke and the occurrence rate of systemic embolism during the duration of the study
Quality of life score | 12 months
  Assessment of the quality of life of patients using a scoring questionnaire adapted to the living conditions of the Algerian population.
  The scoring varies between the lowest score of 12 and highest of 48. Change in quality of life score during the follow-up period will be evaluated by comparing the mean values.

CONTACTS AND LOCATIONS:
Overall Officials: Pr Aoudia Yazid, Principal Investigator — EPH Tipaza; Pr ADJEROUD Naima, Study Chair — Faculty of Medicine of Algiers
Locations (17):
- Algeria (17):
  - Boumaaza Private healthcare, Algiers
  - CHU Mustapha, Algiers
  - BEDAI private healthcare, Annaba
  - Berboucha, Annaba
  - Boudjelal private healthcare, Batna City
  - OKBI Private healthcare, Biskra
  - KHAITER Private healthcare, Blida
  - AOUICHE private healthcare, Constantine
  - HAMDI private healthcare, Constantine
  - Mouffok private healthcare, M'Sila
  - Ali Lahmar private healthcare, Oran
  - CHU Oran, Oran
  - EID private healthcare, Oran
  - Sebbagh Private Healthcare, Sidi Bel Abbes
  - EPH Tipaza, Tipasa
  - Fernane private healthcare, Tizi Ouzou
  - NASSOUR private healthcare, Tlemcen

IPD SHARING:
Plan to Share IPD: No